CLINICAL TRIAL: NCT03975712
Title: Evaluation of the Pravalence of Rathke's Cleft Cyst of Children Under 15 Years
Acronym: PREVA-KPR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: CHU de Besançon
Record Dates: First submitted 2019-05-27; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Rathke's Cleft Cyst
MeSH Terms: conditions — Central Nervous System Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable, no intervention — Not applicable, no intervention

SUMMARY:
The goal of the study was to evaluate the pravalence of Rathke's Cleft Cyst of children under 15 years of age and demonstrate that their prevalence is higher than for patients over 15 years of age, due to their embryonic origin. It is also aimed to describe their aspect on MRI and evaluate the interobserver agreement in the detection of Rathke's Cleft Cyst.

DETAILED DESCRIPTION:
Rathke's cleft cysts (RCC) are benign cystic lesions in the sellar region and correspond to embryonic remnants of the Rathke's pouch. The prevalence of RCC in the literature is higher in adults than in children, but the data for children is limited and outdated. The hypothesis is that the frequency of RCC has been underestimated in children and that it actually decreases with age, especially in adults. The main objective of this descriptive study is to study the prevalence and signal of RCC in children under 15 years of age.

460 encephalic MRIs of children under 15 years of age comprising at least one sagittal sequence without T1-weighted injection and/or a T2 sagittal sequence adapted to the study of the pituitary gland, were analyzed retrospectively. Examination analyses was performed blindly by two radiologists for serous RCC, hypersignal on T2-weighted and isosignal T1-weighted sequences, and mucosal RCC, hyposignal on T2-weighted sequences and hyper or isosignal on T1-weighted sequences. The results were consensually read in case of disagreement on the presence or absence of an RCC.

Of the 460 patients included, the prevalence of RCC was 3% (14/460). 21% of the RCC cases (3/14) were serous and 79% (11/14) were mucosal. Of the 14 patients with RCC, a post-pituitary cyst was also found. The interobserver agreement was strong with a Cohen kappa coefficient of 0.85.

The prevalence of RCC in children under 15 years of age (3%) is higher than that described in the literature (1.2%) and is close to that of adults (3.9%). RCCs are thus intra-sellar lesions of relatively frequent discovery in children, i.e. to identify in order to not erroneously lead to a differential diagnosis including tumors which would lead to a different prognosis, management, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* children aged 15 or under at the time that an MRI was performed exploring the sellar region
* MRI with at least T1 spin echo (SE) sagittal slices with a slice thickness of 2.5 or 3 mm with inter-slice spacing of 0.3 mm and T2 SE with a slice thickness of 2 mm and inter-slice spacing of 0.2 mm.

Exclusion Criteria:

* Patients with incomplete MRI protocol
* Patients whose MRI images had artifacts (patient movement, presence of dental material)
* Patients with suspected pituitary pathology due to endocrine symptomatology (growth retardation, puberty delay, diabetes insipidus) that could be attributed to an intrasellar injury were also excluded.

Age Groups: Child, Adult, Older Adult
Study Population: children aged 15 or under at the time that an MRI was performed exploring the sellar region
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of a strictly intra-pituitary cystic lesion which localization and signal was compatible with an RCC, which type was defined according to its signal | All MRI performed on a period of one year in children under 15 years will be taken into account

SECONDARY OUTCOMES:
Maximum anteroposterior diameter (parallel to the bi-callous plane) of the cyst measured in sagittal section | All MRI performed on a period of one year in children under 15 years will be taken into account
Cyst signal on T2-weighted spin echo sequence compared to cerebrospinal fluid (hypo / iso / hyper signal) and T1-weighted compared to cerebral white matter (hypo / iso / hyper signal) | All MRI performed on a period of one year in children under 15 years will be taken into account
Motive for which brain MRI was performed | All MRI performed on a period of one year in children under 15 years will be taken into account
  The motive can be:
  * benign tumoral pathology
  * neurological manifestations
  * traumatic pathologies
  * other pathologies (deterioration of the general state, exophthalmia).
Dimensions of pituitary | All MRI performed on a period of one year in children under 15 years will be taken into account

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No